CLINICAL TRIAL: NCT01033383
Title: Pilot Study: Dosing Study of Cranberry Capsules for the Prevention of Bacteriuria in Nursing Home Residents
Brief Title: Dosing Study of Cranberry Capsules for the Prevention of Bacteriuria in Nursing Home Residents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0908005581; K23AG028691-01A2 (NIH); UL1RR024139 (NIH); KL2RR024138 (NIH)
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Results first posted 2013-08-15 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-07

CONDITIONS: Bacteriuria
MeSH Terms: conditions — Bacteriuria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 3 placebo capsules (Placebo Comparator): 3 placebo capsules qd
  Interventions: Dietary Supplement: Placebo
- 1 cranberry capsule & 2 placebo capsules (Experimental): 1 active cranberry capsule and 2 placebo capsules qd
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Cranberry Capsule
- 2 cranberry capsules & 1 placebo capsule (Experimental): 2 active cranberry capsules and 1 placebo capsules qd
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Cranberry Capsule
- 3 cranberry capsules (Experimental): 3 active cranberry capsules qd
  Interventions: Dietary Supplement: Cranberry Capsule

INTERVENTIONS:
Dietary Supplement: Placebo — 36 milligram (mg) placebo capsule taken before quiet hours of sleep (qhs).
  Arms: 1 cranberry capsule & 2 placebo capsules; 2 cranberry capsules & 1 placebo capsule; 3 placebo capsules
Dietary Supplement: Cranberry Capsule — 36 milligram (mg) cranberry capsule, taken before quiet hours of sleep (qhs).
  Other Names: Ellura
  Arms: 1 cranberry capsule & 2 placebo capsules; 2 cranberry capsules & 1 placebo capsule; 3 cranberry capsules

SUMMARY:
This study will investigate whether there is a particular dose of cranberry capsules that is effective in preventing the occurrence of urinary tract infections in females at least 65 years of age or older who live in a nursing home and who have a history of urinary tract infections. The Yale research team will be enrolling 80 subjects in total over several nursing home locations within Connecticut.

DETAILED DESCRIPTION:
Each subject was enrolled after providing a baseline urine specimen. Cranberry/placebo capsules were consumed for 30 days. Urine specimens were obtained weekly for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female nursing home residents 65 years of age or older with history of urinary tract infection within the past year.

Exclusion Criteria:

* residents that are not expected to be in the nursing home for at least one month (i.e., short term rehabilitation, pending discharge, terminal [life expectancy < 1 month]);
* residents who are on chronic suppressive antibiotic or anti-infective (i.e., mandelamine) therapy for recurrent UTI;
* residents with end stage renal disease on dialysis (they do not regularly produce urine);
* residents unable to produce a baseline clean catch urine specimen for collection;
* residents on warfarin therapy because of a potential interaction of warfarin and cranberry juice;
* residents with a history of nephrolithiasis because cranberry may increase the risk of nephrolithiasis.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-12; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Juthani-Mehta, MD, Principal Investigator — Yale University
Locations (14):
- United States (14):
  - Northbridge Health Care Center, Bridgeport, Connecticut
  - Sheriden Woods Health Care Center, Bristol, Connecticut
  - The Carolton Chronic and Convalescent Hospital, Fairfield, Connecticut
  - Glastonbury Health Care Center, Glastonbury, Connecticut
  - Middlesex Health Care Center, Middletown, Connecticut
  - Wadsworth Glen Health Care and Rehabilitation Center, Middletown, Connecticut
  - Beacon Brook Health Care Center, Naugatuck, Connecticut
  - Laurel Ridge Health Care Center, Ridgefield, Connecticut
  - Shady Knoll Health Center, Seymour, Connecticut
  - Litchfield Woods Health Care Center, Torrington, Connecticut
  - Maefair Health Care Center, Trumbull, Connecticut
  - Masonicare Health Center, Wallingford, Connecticut
  - Abbott Terracee Health Center, Waterbury, Connecticut
  - Saint Mary Home, West Hartford, Connecticut

REFERENCES:
- [Result] Bianco L, Perrelli E, Towle V, Van Ness PH, Juthani-Mehta M. Pilot randomized controlled dosing study of cranberry capsules for reduction of bacteriuria plus pyuria in female nursing home residents. J Am Geriatr Soc. 2012 Jun;60(6):1180-1. doi: 10.1111/j.1532-5415.2012.03976.x. No abstract available. PMID 22690994
- [Derived] Williams G, Stothart CI, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Nov 10;11(11):CD001321. doi: 10.1002/14651858.CD001321.pub7. PMID 37947276
- [Derived] Williams G, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Apr 17;4(4):CD001321. doi: 10.1002/14651858.CD001321.pub6. PMID 37068952

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of participants occurred at 11 nursing homes from December 2009 to December 2010.
Pre-assignment Details: Once participants consented, they needed to be able to provide a clean catch urine specimen in order to be enrolled.
Groups:
- 3 Placebo Capsules: 3 placebo capsules qd
  Placebo : Three placebo capsules, each 36mg, qhs
- 1 Cranberry Capsule & 2 Placebo Capsules: 1 active cranberry capsule and 2 placebo capsules qd
  1 cranberry capsule & 2 placebo capsules : 1 36mg cranberry capsule, 2 36mg placebo capsules, all qhs
- 2 Cranberry Capsules & 1 Placebo Capsule: 2 active cranberry capsules and 1 placebo capsule qd
  2 cranberry capsules & 1 placebo capsule : 2 36mg cranberry capsules, 1 placebo capsule, all qhs
- 3 Cranberry Capsules: 3 active cranberry capsules qd
  3 cranberry capsules : 3 36mg cranberry capsules qhs
Period: Overall Study
Arm/Group | 3 Placebo Capsules | 1 Cranberry Capsule & 2 Placebo Capsules | 2 Cranberry Capsules & 1 Placebo Capsule | 3 Cranberry Capsules
Started | 20 | 20 | 20 | 20
Completed | 20 | 20 | 20 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 Placebo Capsules | 1 Cranberry Capsule & 2 Placebo Capsules | 2 Cranberry Capsules & 1 Placebo Capsule | 3 Cranberry Capsules | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 20 | 20 | 20 | 20 | 80
Age Continuous [Mean (Standard Deviation); unit: years] | 88.8 (8) | 88.4 (7) | 88.8 (5) | 90.4 (7) | 89.1 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 20 | 20 | 80
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 20 | 80

OUTCOME MEASURES:

1. Primary Outcome: E.Coli Bacteriuria Plus Pyuria
Description: The number of urine cultures and urinalyses (obtained weekly) found with >100,000 CFU/ml growth of E.coli and >10 WBC.
Time Frame: One month
Population: The analysis population were those with completed labs data.
Measure: Number; unit: urine cultures and urinalyses
Units Other Than Participants: Urine cultures and urinalyses
Arm/Group | 3 Placebo Capsules | 1 Cranberry Capsule & 2 Placebo Capsules | 2 Cranberry Capsules & 1 Placebo Capsule | 3 Cranberry Capsules
Number analyzed (Participants) | 20 | 20 | 20 | 20
Number analyzed (Urine cultures and urinalyses) | 76 | 72 | 77 | 73
urine cultures and urinalyses | 33 | 29 | 23 | 25

2. Secondary Outcome: Other Bacteriuria Plus Pyuria
Description: The number of urine cultures and urinalyses (obtained weekly) found with other bacteriuria plus any white blood cells (WBCs) >100,000 colony that include: Proteus, Klebsiella, Enterococcus, beta-hemolytic Streptococci, viridans Streptococci, and organella morganii, Citrobacter freundii, and coagulase-negative Staphylococcus.
Time Frame: one month
Population: The analysis population were those with completed labs data.
Measure: Number; unit: urine cultures and urinalyses
Units Other Than Participants: Urine cultures and urinalyses
Arm/Group | 3 Placebo Capsules | 1 Cranberry Capsule & 2 Placebo Capsules | 2 Cranberry Capsules & 1 Placebo Capsule | 3 Cranberry Capsules
Number analyzed (Participants) | 20 | 20 | 20 | 20
Number analyzed (Urine cultures and urinalyses) | 76 | 72 | 77 | 73
urine cultures and urinalyses | 5 | 4 | 10 | 12

3. Secondary Outcome: Not Growth
Description: The number of not growth, these include no growth, growth <100,000 CFU/ml, growth >100,000 CFU/ml but no WBCs, and mixed flora.
Time Frame: one month
Population: The analysis population were those with completed labs data.
Measure: Number; unit: urine cultures and urinalyses
Units Other Than Participants: Urine cultures and urinalyses
Arm/Group | 3 Placebo Capsules | 1 Cranberry Capsule & 2 Placebo Capsules | 2 Cranberry Capsules & 1 Placebo Capsule | 3 Cranberry Capsules
Number analyzed (Participants) | 20 | 20 | 20 | 20
Number analyzed (Urine cultures and urinalyses) | 76 | 72 | 77 | 73
urine cultures and urinalyses | 38 | 39 | 44 | 36

ADVERSE EVENTS:
Arm/Group | 3 Placebo Capsules | 1 Cranberry Capsule & 2 Placebo Capsules | 2 Cranberry Capsules & 1 Placebo Capsule | 3 Cranberry Capsules
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Of 320 urine specimens that should have been collected by nursing staff, 302 (94%) urine cultures and 294 (92%) urinalyses were obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes